CLINICAL TRIAL: NCT00635089
Title: An Open-Label Safety and Efficacy Study of Reslizumab (CTx55700) for the Treatment of Pediatric Subjects With Eosinophilic Esophagitis Who Completed Study Res-5-0002
Brief Title: Open-Label Extension Study of Reslizumab in Pediatric Subjects With Eosinophilic Esophagitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ception Therapeutics (Industry)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Res-5-0004
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Results first posted 2017-03-23 (Actual); Last update posted 2017-03-23 (Actual); Status verified 2017-02

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophilic Esophagitis; Cinquil
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — reslizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-Label Reslizumab (Other): Open-label reslizumab intravenous (IV) infusion at an initial dose of 1 mg/kg monthly
  Interventions: Drug: reslizumab

INTERVENTIONS:
Drug: reslizumab
  Other Names: Cinquil™; CEP-38072; CTx55700

SUMMARY:
This study is an open-label study where all subjects will receive active drug, reslizumab. Subjects are able to enter this trial only through completion of study Res-05-0002 (NCT00538434).

The goal of the study is to show longer term safety and efficacy in pediatric subjects who have eosinophilic esophagitis.

DETAILED DESCRIPTION:
Subjects will enter this open-label extension study after completing the placebo-controlled, double-blind study Res-5-0002 (NCT00538434). The end of study visit for Res-05-0002 will serve as the screening visit for this trial.

All subjects will receive reslizumab and be followed by their principal investigators in an unblinded fashion. Visits and administration of reslizumab will be monthly.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Received at least two doses of study drug in Study Res-05-0002 (NCT00538434)
* Did not withdraw from Study Res-05-0002 due to drug related adverse event
* Completed End of Treatment Visit for Study Res-05-0002

Exclusion Criteria:

* Pregnant or nursing females
* Concurrent Immunodeficiency
* Current use of immunosuppressive drugs
* Did not tolerate study drug in Study Res-05-0002

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2008-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, MD, Study Director — Cephalon
Locations (36):
- United States (34):
  - The Children's Hospital of Alabama, Birmingham, Alabama
  - University of Arizona Dept. of Pediatrics, Tucson, Arizona
  - Arkansas Children's Hospital/University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Hospital- Pediatric Gastroenterology, Hayward, California
  - Children'S Hospital of Orange County Pediatric Subspecialty Faculty Division of Allergy and Asthma, Orange, California
  - Pediatric Allergy/Immunology, Palo Alto, California
  - Children's Hospital of San Diego, San Diego, California
  - Denver Childrens At Aurora, Colorado, Aurora, Colorado
  - 1st Allergy and Clinical Research Center, Centennial, Colorado
  - Thomas Jefferson University Medical College, Wilmington, Delaware
  - Children's Center for Digestive Health Care, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Children'S Memorial Hospital Division of Gastroenterology Hepatology & Nutrition, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Tuft's Floating Hospital, Boston, Massachusetts
  - Minnesota Gastroenterology, Plymouth, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Creighton University Medical Center, Omaha, Nebraska
  - Las Vegas Pediatric Gastroenterology Associates, Las Vegas, Nevada
  - South Jersey Pediatric Gastroenterology, Mays Landing, New Jersey
  - Mount Sinai School of Medicine, Pediatrics, New York, New York
  - State University of New York (SUNY), Syracuse, New York
  - Center for Digestive Allergic and Immunologic Diseases, Williamsville, New York
  - Pediatric Allergy and Immunology of Duke Medical Center, Durham, North Carolina
  - Cincinnati Children's, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Greenville Health System, Greenville, South Carolina
  - University of Texas Southwest Medical Center, Dallas, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
  - Children's Pavilion, Richmond, Virginia
  - Carilion Medical Center for Children, Roanoke, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Pediatric Allergy and Immunology, Edmonton, Alberta
  - University of Montreal, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open-Label Reslizumab
Started | 190
Completed >/= 16 Weeks of Study | 181
Completed | 112 (Participants who had not withdrawn at the time of study termination.)
Not Completed | 78
Not completed — Adverse Event | 7
Not completed — Lack of Efficacy | 28
Not completed — Protocol Deviation | 4
Not completed — Lost to Follow-up | 8
Not completed — Other | 31

BASELINE CHARACTERISTICS:
Groups:
- Open-Label Reslizumab: Open-label reslizumab IV infusion at an initial dose of 1 mg/kg monthly
Arm/Group | Open-Label Reslizumab
Number analyzed (Participants) | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.1 (3.97)
Age, Customized [Number; unit: participants]
  5 to 11 years | 81
  12 to 19 years | 109
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 148

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs), Serious AEs, or Discontinuation Due to AEs
Description: An AE was defined as any adverse experience, including side effect, injury, toxicity, sensitivity reaction, intercurrent illness, or sudden death, whether or not it was considered related to the use of study drug. Treatment emergent adverse events were those that started any time after the administration of the first dose of study drug (at baseline of this study) and before the cessation of study drug. Serious adverse events that occurred any time after the administration of the first dose of study drug until 30 days after administration of the last dose of study drug were reported as treatment emergent serious adverse events.
Time Frame: From start of study drug until end of treatment (mean [standard deviation {SD}] duration of treatment was 30.0 [5.89] months)
Population: Three additional participants experiences anaphylactic reactions that were upgraded to serious AEs after database lock. These 3 participants are not included in this table summary.
Measure: Number; unit: participants
Arm/Group | Open-Label Reslizumab
Number analyzed (Participants) | 190
participants
  Any AEs | 177
  Severe AEs | 38
  Treatment-related AEs | 63
  Deaths | 0
  Other Serious AEs | 21
  Withdrawn from study due to AEs | 7

2. Secondary Outcome: Mean Change From Baseline to Endpoint in Peak Esophageal Eosinophil Counts
Description: The mean change from baseline in esophageal eosinophil levels was described at week 16 or early withdrawal (if before week 16), using descriptive statistics. Baseline was defined as the last assessment before the first dose of reslizumab, which was the baseline of the double-blind study (NCT00538434) for patients who received reslizumab in the double blind study or the baseline of the open-label study for patients who received placebo during the double-blind study.
Time Frame: Baseline, Week 16 or early withdrawal (if before Week 16)
Population: Participants with an assessment at Baseline and Week 16 (or early withdrawal).
Measure: Mean (Standard Deviation); unit: eosinophils/high power field (hpf)
Arm/Group | Open-Label Reslizumab
Number analyzed (Participants) | 179
eosinophils/high power field (hpf) | -62.0 (77.97)

3. Primary Outcome: Number of Participants With at Least 1 Potentially Clinically Significant Abnormal Hematology Value
Description: Hematology laboratory tests performed include: hemoglobin, hematocrit, red blood cell count, mean cell volume, mean cell hemoglobin, mean cell hemoglobin concentration, platelet count, white blood cell count, and differential count and percentage (polymorphonuclear leukocytes [neutrophils], lymphocytes, eosinophils, monocytes, basophils, platelets).
Time Frame: From start of study drug until end of treatment (mean [SD] duration of treatment was 30.0 [5.89] months)
Population: Participants with a postbaseline result for hematology tests.
Measure: Number; unit: participants
Arm/Group | Open-Label Reslizumab
Number analyzed (Participants) | 188
participants
  Hemoglobin </= 100 g/L | 1
  Hematocrit < 0.30 L/L | 1
  Leukocytes </= 3*10^9/L | 7
  Neutrophils </= 1*10^9/L | 16
  Platelets </= 75*10^9/L | 3

4. Primary Outcome: Number of Participants With at Least 1 Potentially Clinically Significant Abnormal Serum Chemistry Laboratory Test Results or Urinalysis Abnormality
Description: Serum chemistry laboratory tests performed include: calcium, phosphorus, magnesium, sodium, potassium, chloride, creatinine, glucose [nonfasting], blood urea nitrogen, total cholesterol, uric acid, alanine aminotransferase, aspartate aminotransferase, lactate dehydrogenase, gamma glutamyl transpeptidase, alkaline phosphatase, bicarbonate, creatine kinase, total protein, albumin, total bilirubin, direct bilirubin, indirect bilirubin. Urinalysis tests performed include: protein, glucose, ketones, bilirubin, urobilinogen, nitrite content, pH, specific gravity, white blood cells, microscopic (red blood cells, white blood cells, casts, crystals).
Time Frame: From start of study drug until end of treatment (mean [SD] duration of treatment was 30.0 [5.89] months)
Measure: Number; unit: participants
Arm/Group | Open-Label Reslizumab
Number analyzed (Participants) | 190
participants
  Abnormal Serum Chemistry Laboratory Test Results | 0
  Urinalysis Abnormalities | 0

5. Primary Outcome: Number of Participants With at Least 1 Potentially Clinically Significant Abnormal Vital Signs Value
Description: Low systolic blood pressure: < 90 and decrease (↓) of 30 mm Hg from baseline (BL) (ages 5-18); high systolic blood pressure: > 160 and increase (↑) of 30 mm Hg from BL (age 5-12), > 130 and ↑ of 30 mm Hg from BL (age 13-18). Low diastolic blood pressure: < 45 and ↓ of 12 mm Hg from BL (age 5-12), < 55 and ↓ of 12 mm Hg from BL (age 13-18), < 50 and ↓ of 15 mm Hg from BL; high diastolic blood pressure: > 85 and ↑ of 12 mm Hg from BL (ages 5-18). Low heart rate: < 80 and and ↓ of 30 beats per minute (bpm) from BL (age 5-12), < 60 and and ↓ of 30 bpm from BL (age 13-18), < 50 and and ↓ of 15 bpm from BL (age > 18); high heart rate: > 120 and ↑ of 30 bpm from BL (age 5-12), > 100 and ↑ of 30 bpm from BL (age 13-18), > 100 and ↑ of 15 bpm from BL (age > 18). Low oral body temperature: < 35.8° Celsius (age 5 to >18); high oral body temperature: > 38.1° C and ↑ 2° Celsius from BL (age 5-18).
Time Frame: From start of study drug until end of treatment (mean [SD] duration of treatment was 30.0 [5.89] months)
Measure: Number; unit: participants
Arm/Group | Open-Label Reslizumab
Number analyzed (Participants) | 190
participants
  Low systolic blood pressure | 21
  High systolic blood pressure | 18
  Low diastolic blood pressure | 88
  High diastolic blood pressure | 27
  Low heart rate | 42
  High heart rate | 22
  Low oral temperature | 72
  High oral temperature | 2

6. Primary Outcome: Number of Participants With Newly Diagnosed Physical Examination Abnormalities at Endpoint
Description: HEENT=head, eyes, ears, nose and throat.
Time Frame: From start of study drug until end of treatment (mean [SD] duration of treatment was 30.0 [5.89] months)
Measure: Number; unit: participants
Arm/Group | Open-Label Reslizumab
Number analyzed (Participants) | 190
participants
  General appearance | 0
  HEENT | 7
  Neck/thyroid | 0
  Skin | 4
  Lymph nodes | 0
  Heart | 1
  Chest and lungs | 3
  Neurological cranial nerves | 0
  Neurological strength | 0
  Neurological sensation | 0
  Neurological reflexes | 0
  Other | 9

7. Primary Outcome: Infusion Site Evaluations
Description: The infusion site was assessed before treatment and within 30 minutes after the end of the infusion at each monthly treatment visit (or at early withdrawal if before Week 16). The infusion site was graded according to a 5-point scale as follows: 0=no tenderness at IV site, no erythema, no swelling, no induration, no purulence, no palpable venous cord; 1=tender IV site, no erythema, no swelling, no induration, no purulence, no palpable venous cord; 2=tender IV site with erythema, some degree of swelling, no induration, no purulence, no palpable venous cord; 3=tender IV site with erythema and swelling, with induration or palpable venous cord, no purulence; 4=frank vein thrombosis, along with all signs of grade 3 with purulence; IV may stop running because of thrombosis. After the 16-week visit, formal infusion site evaluations were not continued. However, any infusion site reactions were recorded as adverse events and graded as other adverse events.
Time Frame: Day 0, Weeks 4, 8, 12, 16, endpoint (last visit), any time during study (mean [SD] duration of treatment was 30.0 [5.89] months)
Population: Number of Participants Analyzed= all participants in study (n=190); n=number of participants graded at given time point.
Measure: Number; unit: participants
Groups:
- Grade 0: Participants receiving open-label reslizumab IV infusion at an initial dose of 1 mg/kg monthly with an infusion site evaluation grade 0.
- Grade 1: Participants receiving open-label reslizumab IV infusion at an initial dose of 1 mg/kg monthly with an infusion site evaluation grade 1.
- Grade 2: Participants receiving open-label reslizumab IV infusion at an initial dose of 1 mg/kg monthly with an infusion site evaluation grade 2.
- Grade 3: Participants receiving open-label reslizumab IV infusion at an initial dose of 1 mg/kg monthly with an infusion site evaluation grade 3.
- Grade 4: Participants receiving open-label reslizumab IV infusion at an initial dose of 1 mg/kg monthly with an infusion site evaluation grade 4.
Arm/Group | Grade 0 | Grade 1 | Grade 2 | Grade 3 | Grade 4
Number analyzed (Participants) | 190 | 190 | 190 | 190 | 190
participants
  Day 0; n=190 | 178 | 11 | 1 | 0 | 0
  Week 4; n=188 | 179 | 8 | 1 | 0 | 0
  Week 8; n=184 | 181 | 2 | 1 | 0 | 0
  Week 12; n=181 | 175 | 4 | 1 | 1 | 0
  Week 16; n=159 | 154 | 4 | 1 | 0 | 0
  Endpoint; n=190 | 185 | 4 | 1 | 0 | 0
  Any time; n=190 | 190 | 25 | 3 | 1 | 0

8. Primary Outcome: Therapeutic Classification of Concomitant Medications in at Least 10% of Participants
Description: Number of participants receiving therapeutic classes of concomitant medications.
Time Frame: From start of study drug until end of treatment (mean [SD] duration of treatment was 30.0 [5.89] months)
Measure: Number; unit: participants
Arm/Group | Open-Label Reslizumab
Number analyzed (Participants) | 190
participants
  Any concomitant medication | 176
  Analgesics | 93
  Antibacterials for systemic use | 117
  Antiemetics and antinauseants | 28
  Antihistamines for systemic use | 123
  Antiinflammatory and antirheumatic products | 83
  Antipruritics, including antihistamine,anesthetic | 26
  Antivirals for systemic use | 24
  Corticosteroids for systemic use | 40
  Corticosteroids, dermatological preparations | 27
  Cough and cold preparations | 55
  Drugs for acid-related disorders | 59
  Drugs for obstructive airway diseases | 93
  Laxatives | 26
  Mineral supplements | 20
  Nasal preparations | 73
  Ophthalmologicals | 19
  Psychoanaleptics | 49
  Psycholeptics | 33
  Vaccines | 31
  Vitamins | 36

9. Secondary Outcome: Participant's EoE Predominant Symptoms Over Time
Description: The data from the patient's/parent's eosinophilic esophagitis (EoE) Symptom Assessment were used to assess the shift from baseline in Predominant Symptom Assessment. The predominant symptom of the participant's/parent's EoE Symptom Assessment was selected at the double-blind baseline visit and remained the same throughout this study. Using the EoE Symptom Assessment, the participant/parent or legal guardian rated the severity of the previous week's EoE symptoms as none, mild, moderate, severe, or very severe on a 5-point scale. Only the predominant symptom selected for each participant contributed to the overall analysis of the Predominant Symptom Assessment and the subgroup analyses of individual symptoms. Thus, for the Predominant Symptom Analysis, some patients had dysphagia assessed, while others had either abdominal/chest pain or vomiting/regurgitation assessed.
Time Frame: Every 3 weeks from Day 0 up to Week 42 (mean [SD] duration of treatment was 30.0 [5.89] months)
Population: The statistical analysis plan only specified that data would be summarized/described graphically for visual inspection and cannot be summarized.
Arm/Group | Open-Label Reslizumab
Number analyzed (Participants) | 0

10. Secondary Outcome: Physician's EoE Global Assessment Over Time
Description: The data from the participant's/parent's EoE Symptom Assessment, in combination with other observations, were used by physicians to determine the Physician's EoE Global Assessment. All components of the patient's EoE Symptom Assessment were used by physicians to determine the Physician's EoE Global Assessment.
Time Frame: Every 3 weeks from Day 0 up to Week 42 (mean [SD] duration of treatment was 30.0 [5.89] months)
Population: as for outcome 9
Arm/Group | Open-Label Reslizumab
Number analyzed (Participants) | 0

11. Secondary Outcome: Mean Change From Baseline to Endpoint in Selected Child Health Questionnaire (CHQ) Scores
Description: The Child Health Questionnaire comprises 50 items. Specific items are recoded and/or recalibrated. Raw scores for scales (domains calculated over one or more items) are then calculated following set algorithms. The raw scales are then transformed to 0 to 100 scores, except for Change in Health which remains a 1-5 score. Finally two summary measures are calculated based on weighted combinations of selected scales. The Global Health, Physical Summary Score and Psychosocial Summary Score were summarized. For each, scores range from 0 (higher disease activity) to 100 (lower disease activity); higher scores indicate better health.
Time Frame: Baseline through Endpoint (last visit; mean [SD] duration of treatment was 30.0 [5.89] months)
Population: n=participants with an assessment for the given score at Baseline and Endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Reslizumab
Number analyzed (Participants) | 190
units on a scale
  Global Health; n=181 | 4.6 (20.62)
  Physical Summary Scale; n=170 | 3.7 (9.26)
  Psychosocial Summary Scale; n=170 | 3.1 (8.83)

12. Secondary Outcome: Dietary Question Responses at Endpoint
Description: Number of participants answering that they either maintained or changed their diet from the beginning of the double-blind study (ie, NCT00538434). Additionally, for those participants who answered that they changed their diet from the beginning of the double-blind study (column 2), the number of participants in that group who changed by increasing the consistency of their food ('Increased consistency') and the percentage that changed by eating foods that previously worsened EoE ('Added foods'). (Note that these 2 categories are not mutually exclusive, so that someone could have both increased the consistency of the food they were eating AND also eaten foods that previously worsened their EoE symptoms.)
Time Frame: Study endpoint (mean [SD] duration of treatment was 30.0 [5.89] months)
Population: Number of Participants Analyzed=all participants (n=190). The denominator for follow-up questions is the number of participants responding 'No' to the question "Have you maintained your diet since the beginning of the study?" (n=63).
Measure: Number; unit: participants
Groups:
- Maintained Diet From Beginning of Double-blind Study: Participants receiving open-label reslizumab IV infusion at an initial dose of 1 mg/kg monthly who maintained their diet from the beginning of the double-blind study (NCT00538434).
- Changed Diet From Beginning of Double-blind Study: Participants receiving open-label reslizumab IV infusion at an initial dose of 1 mg/kg monthly who changed their diet from the beginning of the double-blind study (NCT00538434).
- Changed by Increasing Consistency of Food: Participants receiving open-label reslizumab IV infusion at an initial dose of 1 mg/kg monthly who changed their diet from the beginning of the double-blind study (NCT00538434) by increasing the consistency of their food.
- Changed by Eating Foods That Previously Worsened EoE: Participants receiving open-label reslizumab IV infusion at an initial dose of 1 mg/kg monthly who changed their diet from the beginning of the double-blind study (NCT00538434) by eating foods that previously worsened EoE.
Arm/Group | Maintained Diet From Beginning of Double-blind Study | Changed Diet From Beginning of Double-blind Study | Changed by Increasing Consistency of Food | Changed by Eating Foods That Previously Worsened EoE
Number analyzed (Participants) | 190 | 190 | 63 | 63
participants | 124 | 63 | 21 | 46

13. Secondary Outcome: Reslizumab Serum Concentrations
Description: Reslizumab serum concentrations obtained in this study were included in ongoing and separate population pharmacokinetic analyses. The Number of Participants Analyzed reflects the number of participants who had concentrations measured following that dose level. Since some participants started on 1 mg/kg and later increased to 2 mg/kg (and are therefore represented in more than one column), the number of participants in each column add up to a greater number than the total in the overall column, which reflects the total number of participants with measurable concentration data in this study. The number of concentrations summarized for that dose level represents more than one concentration per participant in most cases.
Time Frame: Before treatment (within 3 hours) and after treatment (within 3 hours after end of infusion) for doses at Weeks 8 and 12; within 6 days after either dose at Weeks 8 or 12; 2 to 4 weeks after dose at Weeks 8 or 12; and at premature withdrawal.
Population: Number of participants with measurable concentration data at each dose level and overall.
Measure: Mean (Standard Deviation); unit: µg/mL
Units Other Than Participants: Concentrations
Groups:
- Open-Label Reslizumab: 1 mg/kg: Open-label reslizumab IV infusion at 1 mg/kg monthly
- Open-Label Reslizumab: 2 mg/kg: Open-label reslizumab IV infusion at 2 mg/kg monthly
- Open-Label Reslizumab: 3 mg/kg: Open-label reslizumab IV infusion at 3 mg/kg monthly
- Open-Label Reslizumab: Overall: Open-label reslizumab IV infusion at an initial dose of 1 mg/kg monthly, continued at 1 to 3 mg/kg monthly
Arm/Group | Open-Label Reslizumab: 1 mg/kg | Open-Label Reslizumab: 2 mg/kg | Open-Label Reslizumab: 3 mg/kg | Open-Label Reslizumab: Overall
Number analyzed (Participants) | 162 | 100 | 6 | 179
Number analyzed (Concentrations) | 563 | 348 | 9 | 920
µg/mL | 15.747 (11.293) | 29.507 (20.592) | 41.360 (54.952) | 21.202 (17.684)

14. Secondary Outcome: Number of Participants With >/= 1 Confirmed Positive Value for Anti-drug Antibodies (ADA)
Description: Using a validated enzyme-linked immunosorbent assay (ELISA), the number of participants who had at least 1 confirmed positive value for ADA, either on day 0 after having received reslizumab in the double-blind study Res-05-0002 (NCT00538434) or during the course of the open-label study.
Time Frame: From start of study drug until end of treatment (mean [SD] duration of treatment was 30.0 [5.89] months)
Population: Participants with an assessment.
Measure: Number; unit: participants
Arm/Group | Open-Label Reslizumab
Number analyzed (Participants) | 189
participants | 6

ADVERSE EVENTS:
Time Frame: Day 0 through the end of study. The mean duration of treatment within the open-label extension for all participants was 24.7 months (range, 0.0 to 40.5 months).
Arm/Group | Open-Label Reslizumab
Serious Adverse Events (participants affected / at risk) | 21/190
Other Adverse Events (participants affected / at risk) | 167/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Reslizumab (N=190)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Foreign body trauma (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (3)
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Suicide attempt (Psychiatric disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hospitalisation (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Reslizumab (N=190)
Lymphadenopathy (Blood and lymphatic system disorders) | 17 (18)
Abdominal pain (Gastrointestinal disorders) | 22 (23)
Abdominal pain upper (Gastrointestinal disorders) | 17 (51)
Constipation (Gastrointestinal disorders) | 17 (20)
Diarrhoea (Gastrointestinal disorders) | 25 (38)
Nausea (Gastrointestinal disorders) | 23 (27)
Vomiting (Gastrointestinal disorders) | 27 (37)
Fatigue (General disorders) | 12 (21)
Pyrexia (General disorders) | 29 (41)
Food allergy (Immune system disorders) | 15 (16)
Seasonal allergy (Immune system disorders) | 21 (27)
Bronchitis (Infections and infestations) | 14 (18)
Ear infection (Infections and infestations) | 19 (22)
Gastroenteritis (Infections and infestations) | 15 (23)
Gastroenteritis viral (Infections and infestations) | 30 (37)
Influenza (Infections and infestations) | 37 (40)
Nasopharyngitis (Infections and infestations) | 40 (64)
Otitis media (Infections and infestations) | 10 (12)
Sinusitis (Infections and infestations) | 35 (55)
Upper respiratory tract infection (Infections and infestations) | 45 (82)
Viral infection (Infections and infestations) | 14 (15)
Excoriation (Injury, poisoning and procedural complications) | 12 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (18)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (19)
Dizziness (Nervous system disorders) | 14 (20)
Headache (Nervous system disorders) | 50 (118)
Migraine (Nervous system disorders) | 11 (14)
Asthma (Respiratory, thoracic and mediastinal disorders) | 28 (56)
Cough (Respiratory, thoracic and mediastinal disorders) | 31 (69)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 20 (31)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 53 (85)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Acne (Skin and subcutaneous tissue disorders) | 10 (10)
Rash (Skin and subcutaneous tissue disorders) | 20 (38)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.